CLINICAL TRIAL: NCT02792959
Title: Evaluation of Response to the Neoadjuvant Chemotherapy for Advanced Ovarian Cancer by Multimodal Functional Imaging (Fusion MRI and FDG-PET-CT)
Brief Title: Evaluation of Response to the Neoadjuvant Chemotherapy for Advanced Ovarian Cancer by Multimodal Functional Imaging
Acronym: IMOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Roche Pharma AG (Industry); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IB 2013-03
Record Dates: First submitted 2016-04-26; First posted 2016-06-08 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional imaging (Experimental): A pilot study to evaluate the response to neoadjuvant chemotherapy for advanced ovarian cancer by multimodal functional imaging (Fusion MRI and FDG-PET-CT)
  Interventions: Device: Functional Imaging previous the second course; Device: Functional Imaging previous the surgery

INTERVENTIONS:
Device: Functional Imaging previous the second course — Functional Imaging before and after 1 cycle of chemotherapy treatment, in the previous 4 days before the second course: PET1 and MRI1
Device: Functional Imaging previous the surgery — Functional Imaging after 4 cycles of chemotherapy treatment, in the 3 weeks after the chemotherapy, before the interval surgery: PET4 and MRI4 The RECIST evaluation will be done, usually, by scanner to 4 courses of chemotherapy before the surgery interval

SUMMARY:
This study evaluates the therapeutic response by modern FMRI and PET techniques with the perspective to exploit multimodal data (fusion MRI/PET). The Sponsor would like to optimize the respective performances and to define the early assessment criteria, at the first detox, of the treatment efficacy, with and without antiangiogenic agent.

DETAILED DESCRIPTION:
This study evaluates the therapeutic response by modern FMRI and PET techniques with the perspective to exploit multimodal data (fusion MRI/PET). The Sponsor would like to optimize the respective performances and to define the early assessment criteria, at the first detox, of the treatment efficacy, with and without antiangiogenic agent. It is a single center evaluation of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Epithelial ovarian carcinoma, fallopian tube, or primary peritoneal carcinoma FIGO IIIC-IV histologically confirmed by biopsy and documented stage and untreated
* Pre-treatment abdominopelvic PET-CT and MRI within 4 weeks before neoadjuvant chemotherapy.
* During laparoscopy performed by an experienced surgeon in the treatment of ovarian cancer, patient considered ineligible for tumor cell kill at the outset.
* A life expectancy of greater than three months
* An eligible patient for Paclitaxel and Carboplatine based chemotherapy.
* Membership of a social security scheme
* Patient information and signed, dated written informed consent

Exclusion Criteria:

* Pre-treated using chemotherapy, radiology, or surgery for an ovarian cancer.
* Contraindication to MRI with the injection of contrast product, i.e, the first three months pregnancy, claustrophobia, major allergic antecedents, pacemaker, some surgery clips, some heart valves, cava filter, implanter pumps, cochlear implants, metallic extraneous malter.
* Uncontrolled diabetes
* Pregnancy and nursing
* Other uncontrolled medical conditions as thyroid pathology, neuropsychiatric disease, infection, coronary insufficiency or grade 3 - 4 heart disease established by association "New York Heart"
* Patient deprived of liberty and legally protect adult, or not in position to give consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08; Primary Completion 2017-01 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure CAZEAU, MD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Registre des essais cliniques de l'Institut National du Cancer — https://www.e-cancer.fr/Professionnels-de-sante/Le-registre-des-essais-cliniques/Le-registre-des-essais-cliniques
- See also: Site internet du promoteur, l'Institut Bergonié — https://www.bergonie.fr/essais_cliniques/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first steering committee (which met on 30th June, 2015) decided that one patient was not assessable for primary endpoint and had to be replaced. This patient deceased after the first line chemotherapy.
Period: Overall Study
Arm/Group | Functional Imaging
Started | 11
Completed | 10
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Functional Imaging
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 67.0 [41.8 to 77.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Proven epithelial carcinoma of gynaecological origin [Count of Participants; unit: Participants]
  Yes | 11
  No | 0
Location of the tumour [Count of Participants; unit: Participants]
  Ovaries | 9
  Trunk | 1
  Primitive peritoneal | 1
Histological type [Count of Participants; unit: Participants]
  Serous | 11
  Other type | 0
Stage of the tumour [Count of Participants; unit: Participants] — The stage of tumour is graded from I-a to IV-c. The higher the stage number/letter is, the further the cancer has spread.
  Participants
    III-c | 5
    IV | 6
Total Fagotti Score [Count of Participants; unit: Participants] — The Fagotti score ranges from 0 to 14 and is used to evaluate the peritoneal damage of patients. This score was collected during pretherapy. The higher the stage number is, the further the cancer has spread.
  The Fagotti questionnaire has 7 items. A subscale value of 0 or 2 is assigned depending on whether the disease is present in those specific sites : large omentum, peritoneal carcinosis , diaphragmatic carcinosis, mesenteric retraction, intestinal infiltration, stomach infiltration,liver metastases.
  The sum of all subscale values corresponds to Fagotti score.
  Participants
    4 | 2
    8 | 4
    10 | 3
    12 | 1
    Not available | 1
Performance status ECOG [Count of Participants; unit: Participants] — Performance status ECOG questionnaire is a tool for measuring the degree of autonomy of a person through his or her ability to carry out certain tasks of daily life.
  The score ranges from 0 (able to carry out the same activity as before the illness without any restrictions) and stage 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) to stade 4 (unable to take care of himself, bedridden or in a chair all the time).
  Participants
    Not available | 1
    0 | 4
    1 | 6
Weight [Median (Full Range); unit: Kg] | 59.0 [54.0 to 78.0]
Height [Median (Full Range); unit: cm] | 164.0 [150.0 to 173.0]
Number of measurable initial lesions [Count of Participants; unit: Participants]
  1 | 2
  2 | 2
  3 | 1
  4 | 3
  5 | 3
Number of non-target lesions [Count of Participants; unit: Participants]
  2 | 3
  3 | 5
  4 | 1
  5 | 2
Sum of the diameters [Median (Full Range); unit: diameters] | 176.0 [70.0 to 310.0]

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Individual Intra-class Correlation Coefficients by Location
Description: Individual intra-class correlation coefficients by location (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter SUVmax of functional imaging positron emission tomography. The functional imaging positron emission tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: Pre-therapeutic
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.992 [0.969 to 0.998]
  Sus-mesocolic | 0.997 [0.987 to 0.999]
  Sub-mesocolic | 0.983 [0.937 to 0.996]
  Pelvis | 0.997 [0.988 to 0.999]
  Viscera | 0.951 [0.826 to 0.987]
  ADP | 0.960 [0.853 to 0.990]

2. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Average Intra-class Correlation Coefficients by Location
Description: Average intra-class correlation coefficients(Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter SUVmax of functional imaging positron emission tomography.
  The functional imaging positron emission tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: Pre-therapeutic
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.996 [0.984 to 0.999]
  Sus-mesocolic | 0.999 [0.993 to 1.000]
  Sub-mesocolic | 0.992 [0.968 to 0.998]
  Pelvis | 0.998 [0.994 to 1.000]
  Viscera | 0.975 [0.905 to 0.994]
  ADP | 0.980 [0.921 to 0.995]

3. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Individual Intra-class Correlation Coefficients by Location
Description: Individual intra-class correlation coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter MTV of functional imaging Positron Emission Tomography.
  The functional imaging positron emission tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: Pre-therapeutic
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.482 [-0.079 to 0.833]
  Sus-mesocolic | 0.450 [-0.165 to 0.824]
  Sub-mesocolic | 0.137 [-0.606 to 0.698]
  Pelvis | 0.747 [0.298 to 0.929]
  Viscera | 0.023 [-0.586 to 0.616]
  ADP | 0.881 [0.614 to 0.969]

4. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Average Intra-class Correlation Coefficients by Location
Description: Average intra-class correlation coefficients (Absolute agreement) arepresented by location to evaluate the reliability between observers of quantization parameter MTV of functional imaging Positron Emission Tomography.
  The functional imaging Positron Emission Tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: Pre-therapeutic
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.650 [-0.173 to 0.909]
  Sus-mesocolic | 0.621 [-0.396 to 0.904]
  Sub-mesocolic | 0.241 [-3.081 to 0.822]
  Pelvis | 0.855 [0.460 to 0.963]
  Viscera | 0.044 [-2.827 to 0.762]
  ADP | 0.937 [0.761 to 0.984]

5. Primary Outcome: Inter-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter ADC of functional imaging Magnetic Resonance Imaging.
  The Magnetic Resonance Imaging will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: Pretherapeutic
Population: For patients with lesions by location at baseline : only eight patients had supra-diaphragmatic lesions and nine had ADP lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.813 [0.292 to 0.960]
  Sus-mesocolic | 0.922 [0.723 to 0.980]
  Sub-mesocolic | 0.794 [0.393 to 0.944]
  Pelvis | 0.178 [-0.567 to 0.718]
  Viscera | 0.983 [0.925 to 0.996]
  ADP: number analyzed (Participants) | 9
  ADP | 0.974 [0.896 to 0.994]

6. Primary Outcome: Inter-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Average Intra-class Correlation Coefficients by Location
Description: Average intra-class correlation coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter ADC of functional imaging Magnetic Resonance Imaging.
  The Magnetic Resonance Imaging will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: Pretherapeutic
Population: For patients with lesions by location at baseline: only eight patients had supra-diaphragmatic lesions and nine had ADP lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.897 [0.452 to 0.980]
  Sus-mesocolic | 0.960 [0.834 to 0.990]
  Sub-mesocolic | 0.885 [0.564 to 0.971]
  Pelvis | 0.302 [-2.620 to 0.836]
  Viscera | 0.991 [0.961 to 0.998]
  ADP: number analyzed (Participants) | 9
  ADP | 0.987 [0.945 to 0.997]

7. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation (Absolute agreement) are presented by location to evaluate the reliability within observers of quantization parameter SUVmax of functional imaging Positron Emission Tomography (PET).
  The functional imaging Positron Emission Tomography (PET) will be interpreted twice by radiologist and nuclear medicine specialist.
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.992 [0.969 to 0.998]
  Sus-mesocolic | 0.884 [0.607 to 0.970]
  Sub-mesocolic | 0.983 [0.934 to 0.996]
  Pelvis | 0.998 [0.993 to 1.000]
  Viscera | 0.317 [-0.332 to 0.770]
  ADP | 0.977 [0.913 to 0.994]

8. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter SUVmax of functional imaging Positron Emission Tomography (PET) .
  The functional imaging Positron Emission Tomography (PET) will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.996 [0.684 to 0.999]
  Sus-mesocolic | 0.938 [0.755 to 0.985]
  Sub-mesocolic | 0.991 [0.966 to 0.998]
  Pelvis | 0.999 [0.996 to 1.000]
  Viscera | 0.482 [-0.993 to 0.870]
  ADP | 0.989 [0.954 to 0.997]

9. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Individual Intra-class Correlation Coefficients by Location
Description: Individual intra-class correlation coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter MTV of functional imaging Positron Emission Tomography (PET).
  The functional imaging Positron Emission Tomography (PET) will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After one cycle of chemoterapy, 3 weeks
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.504 [-0.537 to 0.842]
  Sus-mesocolic | 0.882 [0.618 to 0.969]
  Sub-mesocolic | 0.210 [-0.439 to 0.719]
  Pelvis | 0.699 [0.200 to 0.915]
  Viscera | 0.486 [-0.137 to 0.840]
  ADP | 0.994 [0.976 to 0.998]

10. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Average Intra-class Correlation Coefficients by Location
Description: as for outcome 9
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.670 [-0.114 to 0.914]
  Sus-mesocolic | 0.937 [0.764 to 0.984]
  Sub-mesocolic | 0.347 [-1.564 to 0.837]
  Pelvis | 0.823 [0.333 to 0.955]
  Viscera | 0.654 [-0.318 to 0.913]
  ADP | 0.997 [0.988 to 0.999]

11. Primary Outcome: Inter-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter ADC of Magnetic Resonance Imaging (MRI).
  The Magnetic Resonance Imaging will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: For patients with lesions by location after one cycle of chemotherapy : only eight patients had supra-diaphragmatic lesions and nine had ADP lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.807 [0.321 to 0.958]
  Sus-mesocolic | 0.340 [-0.154 to 0.757]
  Sub-mesocolic | -0.080 [-0.703 to 0.564]
  Pelvis | 0.566 [-0.055 to 0.871]
  Viscera | 0.747 [0.240 to 0.931]
  ADP: number analyzed (Participants) | 9
  ADP | 0.863 [0.537 to 0.967]

12. Primary Outcome: Inter-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Average Intra-class Correlation Coefficients by Location
Description: Average intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter ADC of Magnetic Resonance Imaging (MRI).
  The Magnetic Resonance Imaging will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: For patients with lesions by location after once cycle of chemotherapy: only eight patients had supra-diaphragmatic lesions and nine had ADP lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.893 [0.486 to 0.978]
  Sus-mesocolic | 0.507 [-0.365 to 0.862]
  Sub-mesocolic | 0.885 [0.564 to 0.971]
  Pelvis | 0.723 [-0.116 to 0.931]
  Viscera | 0.855 [0.387 to 0.964]
  ADP: number analyzed (Participants) | 9
  ADP | 0.926 [0.698 to 0.983]

13. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter SUVmax of functional imaging positron emission tomography (PET) .
  The functional imaging positron emission tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: For patients with lesions by location after four cycles of chemotherapy: No patients with lesions in supra-diaphragmatic and viscera locations
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 0
  Sus-mesocolic | 0.923 [0.738 to 0.980]
  Sub-mesocolic | 0.953 [0.824 to 0.988]
  Pelvis | 0.962 [0.856 to 0.990]
  Viscera: number analyzed (Participants) | 0
  ADP | 0.942 [0.796 to 0.985]

14. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter SUVmax of functional imaging positron emission tomography (PET).
  The functional imaging positron emission tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 0
  Sus-mesocolic | 0.960 [0.849 to 0.990]
  Sub-mesocolic | 0.976 [0.904 to 0.994]
  Pelvis | 0.981 [0.922 to 0.995]
  Viscera: number analyzed (Participants) | 0
  ADP | 0.970 [0.887 to 0.992]

15. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter MTV of functional imaging Positron Emission Tomography (MTV).
  The functional imaging Positron Emission Tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After four cycles of chemoterapy, 12 weeks
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 0
  Sus-mesocolic | 0.957 [0.838 to 0.989]
  Sub-mesocolic | 0.248 [-0.368 to 0.733]
  Pelvis | 0.998 [0.992 to 0.999]
  Viscera: number analyzed (Participants) | 0
  ADP | 0.943 [0.794 to 0.986]

16. Primary Outcome: Inter-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - AverageIntra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter MTV of functional imaging Positron Emission Tomography (PET).
  The functional imaging Positron Emission Tomography will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 0
  Sus-mesocolic | 0.978 [0.912 to 0.995]
  Sub-mesocolic | 0.398 [-1.163 to 0.846]
  Pelvis | 0.999 [0.996 to 1.000]
  Viscera: number analyzed (Participants) | 0
  ADP | 0.971 [0.885 to 0.993]

17. Primary Outcome: Inter-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter ADC of functional imaging Magnetic Resonance Imaging (MRI).
  The Magnetic Resonance Imaging will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: For patients with lesions by location after four cycles of chemotherapy: only eight patients had supra-diaphragmatic lesions (or ADP lesions).
Measure: Number (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.961 [0.804 to 0.992]
  Sus-mesocolic | 0.730 [0.265 to 0.924]
  Sub-mesocolic | 0.862 [0.543 to 0.964]
  Pelvis | 0.543 [0.059 to 0.861]
  Viscera | 0.834 [0.491 to 0.955]
  ADP: number analyzed (Participants) | 8
  ADP | 1.000 [1.000 to 1.000]

18. Primary Outcome: Inter-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability between observers of quantization parameter of ADC functional imaging Magnetic Resonance Imaging (MRI).
  The Magnetic Resonance Imaging will be interpreted independently by 2 radiologists and 2 nuclear medicine specialists, in blind to results found by the other.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.980 [0.891 to 0.996]
  Sus-mesocolic | 0.844 [0.419 to 0.960]
  Sub-mesocolic | 0.926 [0.704 to 0.982]
  Pelvis | 0.703 [0.126 to 0.925]
  Viscera | 0.910 [0.659 to 0.977]
  ADP: number analyzed (Participants) | 8
  ADP | 1.000 [1.000 to 1.000]

19. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter ADC of functional imaging positron emission tomography (PET).
  The functional imaging positron emission tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: Pre-therapeutic
Population: For patients with lesions by location at baseline: only one patient with lesions in viscera locations
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 1.000 [1.000 to 1.000]
  Sus-mesocolic | 0.998 [0.991 to 0.999]
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 1.000 [0.998 to 1.000]
  Pelvis | 0.997 [0.987 to 0.999]
  Viscera: number analyzed (Participants) | 1
  Viscera | 1.000
  ADP | 0.985 [0.942 to 0.996]

20. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter SUVmax of functional imaging positron emission tomography (PET) .
  The imaging positron emission tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: Pre-therapeutic
Population: For patients with lesions by location at baseline: only one patients with lesions in viscera locations and nine patients with sus-mesocolic lesion
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 1.000 [1.000 to 1.000]
  Sus-mesocolic | 0.999 [0.995 to 1.000]
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 1.000 [0.999 to 1.000]
  Pelvis | 0.998 [0.994 to 1.000]
  Viscera: number analyzed (Participants) | 1
  Viscera | 1.000
  ADP | 0.992 [0.970 to 0.998]

21. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameters functional imaging Positron Emission Tomography (MTV).
  The functional imaging Positron Emission Tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: Pre-therapeutic
Population: For patients with lesions by location at baseline : only nine patients with sub-mesocolic lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.987 [0.951 to 0.997]
  Sus-mesocolic | 0.622 [0.041 to 0.890]
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 0.493 [-0.212 to 0.858]
  Pelvis | 0.847 [0.513 to 0.959]
  Viscera | 0.042 [-0.572 to 0.623]
  ADP | 0.934 [0.770 to 0.983]

22. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients by Location (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameters MTV of functional imaging Positron Emission Tomography.
  The functional imaging Positron Emission Tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: Pre-therapeutic
Population: For patients with lesions by location at baseline : only nine patients with sub-mesocolic lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.993 [0.975 to 0.998]
  Sus-mesocolic | 0.767 [0.079 to 0.942]
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 0.660 [-0.538 to 0.924]
  Pelvis | 0.917 [0.678 to 0.979]
  Viscera | 0.080 [-2.668 to 0.771]
  ADP | 0.966 [0.870 to 0.991]

23. Primary Outcome: Intra-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observers of quantization parameter ADC of Magnetic Resonance Imaging (MRI).
  The Magnetic Resonance Imaging will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: Pretherapeutic
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.747 [0.136 to 0.944]
  Sus-mesocolic | 0.894 [0.634 to 0.972]
  Sub-mesocolic | 0.452 [-0.122 to 0.821]
  Pelvis | 0.217 [-0.481 to 0.730]
  Viscera | 0.639 [0.093 to 0.895]
  ADP: number analyzed (Participants) | 9
  ADP | 0.961 [0.839 to 0.991]

24. Primary Outcome: Intra-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observers of quantization parameter ADC of Magnetic Resonance Imaging (MRI) .
  The Magnetic Resonance Imaging will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: Pretherapeutic
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.855 [0.240 to 0.971]
  Sus-mesocolic | 0.944 [0.776 to 0.986]
  Sub-mesocolic | 0.623 [-0.279 to 0.902]
  Pelvis | 0.356 [-1.855 to 0.844]
  Viscera | 0.780 [0.170 to 0.944]
  ADP: number analyzed (Participants) | 9
  ADP | 0.980 [0.912 to 0.995]

25. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter SUV max of functional imaging positron emission tomography (PET).
  The functional imaging positron emission tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After one cycle of chemoterapy, 3 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.893 [0.636 to 0.972]
  Sus-mesocolic | 0.998 [0.994 to 1.000]
  Sub-mesocolic | 0.993 [0.970 to 0.998]
  Pelvis | 0.997 [0.987 to 0.999]
  Viscera | 0.317 [-0.332 to 0.770]
  ADP | 1.000 [1.000 to 1.000]

26. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter SUVmax of functional imaging positron emission tomography (PET).
  The functional imaging positron emission tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After once cycle of chemoterapy, 3 weeks
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.943 [0.777 to 0.986]
  Sus-mesocolic | 0.999 [0.997 to 1.000]
  Sub-mesocolic | 0.996 [0.985 to 0.999]
  Pelvis | 0.999 [0.994 to 1.000]
  Viscera | 0.482 [-0.993 to 0.870]
  ADP | 0.482 [-0.993 to 0.870]

27. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter MTV of functional imaging Positron Emission Tomography (PET).
  The functional imaging Positron Emission Tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After one cycle of chemoterapy, 3 weeks
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.789 [0.384 to 0.942]
  Sus-mesocolic | 0.898 [0.661 to 0.973]
  Sub-mesocolic | 0.967 [0.866 to 0.992]
  Pelvis | 0.329 [-0.311 to 0.774]
  Viscera | 0.193 [-0.450 to 0.710]
  ADP | 0.997 [0.988 to 0.999]

28. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter MTV of functional imaging Positron Emission Tomography (PET).
  The functional imaging Positron Emission Tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After once cycle of chemotherapy, 3 weeks
Population: Eligible and evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 0.882 [0.555 to 0.970]
  Sus-mesocolic | 0.946 [0.796 to 0.986]
  Sub-mesocolic | 0.983 [0.928 to 0.996]
  Pelvis | 0.495 [-0.903 to 0.873]
  Viscera | 0.323 [-1.634 to 0.830]
  ADP | 0.999 [0.994 to 1.000]

29. Primary Outcome: Intra-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Individual Intra-class Correlation Coefficients by Location
Description: as for outcome 23
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: For patients with lesions by location after one cycle of chemotherapy: only eight patients had supra-diaphragmatic lesions and nine had ADP lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.607 [-0.155 to 0.909]
  Sus-mesocolic | 0.613 [0.038 to 0.887]
  Sub-mesocolic | -0.043 [-0.739 to 0.600]
  Pelvis | 0.451 [-0.177 to 0.826]
  Viscera | 0.792 [0.392 to 0.943]
  ADP: number analyzed (Participants) | 9
  ADP | 0.996 [0.984 to 0.999]

30. Primary Outcome: Intra-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observers of quantization parameter ADC of Magnetic Resonance Imaging (MRI).
  The Magnetic Resonance Imaging will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: as for outcome 29
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.755 [-0.368 to 0.952]
  Sus-mesocolic | 0.760 [0.074 to 0.940]
  Sub-mesocolic | -0.091 [-5.666 to 0.750]
  Pelvis | 0.622 [-0.429 to 0.905]
  Viscera | 0.884 [0.563 to 0.971]
  ADP: number analyzed (Participants) | 9
  ADP | 0.998 [0.992 to 1.000]

31. Primary Outcome: Individual Intra-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter SUVmax of functional imaging positron emission tomography (PET).
  The functional imaging positron emission tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After four cycles of chemoterapy, 12 weeks
Population: For patients with lesions by location after one cycle of chemotherapy: only one patients had sus-mesocolic lesions, nine sub-mesocolic lesion, one ADP lesions and no patient had visceral lesion.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic | 1.000 [1.000 to 1.000]
  Sus-mesocolic: number analyzed (Participants) | 1
  Sus-mesocolic | 1.000
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 1.000 [0.999 to 1.000]
  Pelvis | 0.971 [0.891 to 0.993]
  Viscera: number analyzed (Participants) | 0
  ADP: number analyzed (Participants) | 1
  ADP | 1.000

32. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Maximum Standardized Uptake Value (SUVmax) - Average Intra-class Correlation Coefficients by Location
Description: as for outcome 26
Time Frame: After four cycles of chemoterapy, 12 weeks
Population: Eligible and evaluable population. Only one patient had sus-mesocolic lesions, one patient ADP lesions, nine patients sub-mesocolic lesions and no patient had supra-diaphragmatic or viscera lesions
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 0
  Sus-mesocolic: number analyzed (Participants) | 1
  Sus-mesocolic | 1.000
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 1.000 [0.998 to 1.000]
  Pelvis | 0.944 [0.803 to 0.986]
  Viscera: number analyzed (Participants) | 0
  ADP: number analyzed (Participants) | 1
  ADP | 1.000

33. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter MTV functional imaging positron emission tomography (PET).
  The functional imaging positron emission tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After four cycle of chemoterapy, 12 weeks
Population: For patients with lesions by location after four cycles of chemotherapy: No patients with lesions in the location of supra-diaphragmatic and viscera
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 0
  Sus-mesocolic | 0.794 [0.385 to 0.944]
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 0.794 [0.322 to 0.950]
  Pelvis | 0.975 [0.908 to 0.994]
  Viscera: number analyzed (Participants) | 0
  ADP | 0.987 [0.950 to 0.997]

34. Primary Outcome: Intra-rater Reliability of Positron Emission Tomography (PET) Metabolic Tumoral Volume (MTV) - Average Intra-class Correlation Coefficients by Location
Description: Average Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observer of quantization parameter MTV functional imaging positron emission tomography (PET).
  The functional imaging positron emission tomography will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: For patients with lesions by location after four cycles of chemotherapy: No patients with supra-diaphragmatic lesions or viscera lesions.
Measure: Number (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 0
  Sus-mesocolic | 0.885 [0.556 to 0.971]
  Sub-mesocolic: number analyzed (Participants) | 9
  Sub-mesocolic | 0.885 [0.487 to 0.974]
  Pelvis | 0.987 [0.952 to 0.997]
  Viscera: number analyzed (Participants) | 0
  ADP | 0.993 [0.974 to 0.998]

35. Primary Outcome: Intra-rater Reliability of Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Individual Intra-class Correlation Coefficients by Location
Description: Individual Intra-class Correlation Coefficients (Absolute agreement) are presented by location to evaluate the reliability within observers of quantization parameter ADC of functional imaging Magnetic Resonance Imaging (MRI).
  The Magnetic Resonance Imaging will be interpreted independently twice by the same radiologist and nuclear medicine specialist.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: For patients with lesions (by location) after four cycles of chemotherapy: only eight patients had supra-diaphragmatic lesions (or ADP lesions) and nine had sus-mesocolic lesions.
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.930 [0.703 to 0.986]
  Sus-mesocolic: number analyzed (Participants) | 9
  Sus-mesocolic | 0.654 [0.038 to 0.910]
  Sub-mesocolic | 0.767 [0.302 to 0.937]
  Pelvis | 0.088 [-0.467 to 0.639]
  Viscera | 0.686 [0.184 to 0.910]
  ADP: number analyzed (Participants) | 8
  ADP | 0.804 [0.320 to 0.957]

36. Primary Outcome: Intra-rater Reliability of PET Magnetic Resonance Imaging (MRI) Apparent Diffusion Coefficient (ADC) - Average Intra-class Correlation Coefficients by Location
Description: as for outcome 30
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: as for outcome 35
Measure: Geometric Mean (95% Confidence Interval); unit: proportion of agreement
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
proportion of agreement
  Supra-diaphragmatic: number analyzed (Participants) | 8
  Supra-diaphragmatic | 0.964 [0.826 to 0.993]
  Sus-mesocolic: number analyzed (Participants) | 9
  Sus-mesocolic | 0.791 [0.073 to 0.953]
  Sub-mesocolic | 0.868 [0.463 to 0.967]
  Pelvis | 0.162 [-1.753 to 0.780]
  Viscera | 0.814 [0.311 to 0.953]
  ADP: number analyzed (Participants) | 8
  ADP | 0.891 [0.485 to 0.978]

37. Secondary Outcome: Spearman Correlation Coefficient Between Marker CA125 and the Relative Variations (Between Pretherapeutic and After One Cycle of Chemotherapy) of the PET Parameters (SUVmax, MTV, SUVN, SUL and TLG)
Description: In this section, only the maximum values of the PET parameters (SUVmax, MTV, SUVN, SUL, TLG) and the minimum values of the MRI parameters (ADC) of each patient were taken into account for all lesions present at each evaluation time (pre-therapy, after 1 cycle of chemotherapy, after 4 cycles of chemotherapy). In other words, without paying attention to assessment times and the location of the lesion, for each patient, the highest value of SUVmax, MTV, SUVN, SUL, TLG and the lowest ADC value was taken into account in the analyse.
  The appearance of new lesions (not present at baseline) has not been taken into account in the calculation of relative variations.
  The disappearance of pre-existing lesions at baseline has been taken into account in the calculation of relative variations.
  Relative variations has been calculated as the difference between the values collected after 1 cycle of chemotherapy and the pre-therapeutic value divided by the pre-therapeutic value.
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Eligible and evaluable population
Measure: Number (95% Confidence Interval); unit: Spearman's correlation coefficient
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
Spearman's correlation coefficient
  Spearman correlation test statistics between CA125 and relative variation of PET parameter SUVmax | -0.091 [-0.679 to 0.575]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter MTV | -0.030 [-0.647 to 0.612]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter SUVN | -0.212 [-0.737 to 0.491]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter SUL | -0.212 [-0.737 to 0.491]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter TLG | -0.164 [-0.715 to 0.526]

38. Secondary Outcome: Spearman Correlation Coefficient Between Marker CA125 and the Relative Variations (Between Pre-therapeutic and After Four Cycles of Chemotherapy) of the PET Parameters (SUVmax, MTV, SUVN, SUL and TLG)
Description: In this section, only the maximum values of the PET parameters (SUVmax, MTV, SUVN, SUL, TLG) and the minimum values of the MRI parameters (ADC) of each patient were taken into account for all lesions present at each evaluation time (pre-therapy, after 1 cycle of chemotherapy, after 4 cycles of chemotherapy). In other words, without paying attention to assessment times and the location of the lesion, for each patient, the highest value of SUVmax, MTV, SUVN, SUL, TLG and the lowest ADC value was taken into account in the analyse.
  The appearance of new lesions (not present at baseline) has not been taken into account in the calculation of relative variations.
  The disappearance of pre-existing lesions at baseline has been taken into account in the calculation of relative variations.
  Relative variations has been calculated as the difference between the values collected after 4 cycles of chemotherapy and the pre-therapeutic value divided by the pre-therapeutic value.
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: Eligible and evaluable population
Measure: Number (95% Confidence Interval); unit: Spearman's correlation coefficient
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
Spearman's correlation coefficient
  Spearman correlation test statistics between CA125 and relative variation of PET parameter SUVmax | 0.811 [0.082 to 0.967]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter MTV | 0.775 [-0.012 to 0.960]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter SUVN | 0.811 [0.082 to 0.967]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter SUL | 0.811 [0.082 to 0.967]
  Spearman correlation test statistics between CA125 and relative variation of PET parameter TLG | 0.775 [-0.012 to 0.960]

39. Secondary Outcome: Spearman Correlation Test Between the Relative Variation of Apparent Diffusion Coefficient (ADC) and Marker CA125
Description: In this section, only the maximum values of the PET parameters (SUVmax, MTV, SUVN, SUL, TLG) and the minimum values of the MRI parameters (ADC) of each patient were taken into account for all lesions present at each evaluation time (pre-therapy, after 1 cycle of chemotherapy, after 4 cycles of chemotherapy. In other words, for each patient, the highest value of SUVmax, MTV, SUVN, SUL, TLG and the lowest ADC value was taken into account in the analyses.
  The appearance of new lesions (not present at baseline) has not been taken into account in the calculation of relative variations.
  The disappearance of pre-existing lesions at baseline has been taken into account in the calculation of relative variations.
  Relative variations has been calculated as the difference between the values collected after 1 or 4 cycles of chemotherapy and the pre-therapeutic value divided by the pre-therapeutic value.
Time Frame: After one and four cycle(s) of chemotherapy (after 3 and 12 weeks)
Measure: Number (95% Confidence Interval); unit: Spearman's correlation coefficient
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
Spearman's correlation coefficient
  Relative variations between pre-therapeutic and after one cycle of chemotherapy | 0.103 [-0.567 to 0.685]
  Relative variations between pre-therapeutic and after four cycles of chemotherapy | -0.571 [-0.919 to 0.361]

40. Secondary Outcome: Complete Surgery Resection
Time Frame: Interval surgery visit: up to 3 weeks after cycle 4 of chemotherapy and until the day before the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
Participants
  Yes | 10
  No | 0

41. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter SUVmax by Response as Per RECIST V1.1
Description: In this section, only the maximum values of the PET parameters (SUVmax, MTV, SUVN, SUL, TLG) and the minimum values of the MRI parameters (ADC) of each patient were taken into account for all lesions present at each evaluation time (pre-therapy, after 1 cycle of chemotherapy, after 4 cycles of chemotherapy. In other words, for each patient, the highest value of SUVmax, MTV, SUVN, SUL, TLG and the lowest ADC value was taken into account in the analyses.
  Relative variations has been calculated as the difference between the values collected after 1 or 4 cycles (C1 or C4) of chemotherapy and the pre-therapeutic value (C0) divided by the pre-therapeutic value (C0).
Time Frame: After one cycle of chemotherapy, 3 weeks
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response | -25.4 (33.1)
  Stable disease | -9.6 (29.8)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Non-Inferiority — alpha=5%; p = 0.602, Kruskal-Wallis; Mean Difference (Net) = 0.273

42. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter SUVmax by Response as Per RECIST V1.1
Description: In this section, only the maximum values of the PET parameters (SUVmax, MTV, SUVN, SUL, TLG) and the minimum values of the MRI parameters (ADC) of each patient were taken into account for all lesions present at each evaluation time (pre-therapy, after 1 cycle of chemotherapy, after 4 cycles of chemotherapy. In other words, for each patient, the highest value of SUVmax, MTV, SUVN, SUL, TLG and the lowest ADC value was taken into account in the analyses.
  RRelative variations has been calculated as the difference between the values collected after 1 or 4 cycles (C1 or C4) of chemotherapy and the pre-therapeutic value (C0) divided by the pre-therapeutic value (C0).
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: Relative variations of SUVmax by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -67.3 (29.3)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -11.3 (31.1)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.067, Kruskal-Wallis; Mean Difference (Net) = 3.361

43. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter MTV by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After four cycles of chemotherapy, 12 weeks
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response | -94.7 (11.4)
  Stable disease | 12.9 (52.9)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.036, Kruskal-Wallis; Mean Difference (Net) = 4,390

44. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter MTV by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Relative variations of MTV by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -38.5 (47.6)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -3.3 (5.4)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.296, Kruskal-Wallis; Mean Difference (Net) = 1.091

45. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter SUVN by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Relative variations of SUVN by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -21.8 (28.8)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -15.6 (22.1)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.794, Kruskal-Wallis; Mean Difference (Net) = 0.068

46. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter SUVN by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: Relative variations of SUVN by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -65.2 (29.4)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -16.2 (30.2)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.067, Kruskal-Wallis; Mean Difference (Net) = 3.361

47. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter TLG by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Relative variations of TLG by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -63.5 (52.4)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -15.2 (12.9)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.296, Kruskal-Wallis; Mean Difference (Net) = 1,091

48. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter TLG by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: Relative variations of TLG by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -97.7 (9.4)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -7.5 (18.2)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.036, Kruskal-Wallis; Mean Difference (Net) = 4.390

49. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter SUL by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Relative variations of TLG by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -24.9 (31.9)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -21.8 (11.4)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.794, Kruskal-Wallis; Mean Difference (Net) = 0.068

50. Secondary Outcome: Descriptive Statistics of Relative Variations of PET Parameter SUL by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: Relative variations of TLG by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | -66.9 (29.0)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -14.7 (33.8)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.036, Kruskal-Wallis; Mean Difference (Net) = 4.390

51. Secondary Outcome: Descriptive Statistics of Relative Variations of MRI Parameter ADC by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After one cycle of chemotherapy, 3 weeks
Population: Relative variations of ADC by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | 9.3 (209.7)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | 4.3 (25.1)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.602, Kruskal-Wallis; Mean Difference (Net) = 0.273

52. Secondary Outcome: Descriptive Statistics of Relative Variations of MRI Parameters ADC by Response as Per RECIST V1.1
Description: as for outcome 41
Time Frame: After four cycles of chemotherapy, 12 weeks
Population: Relative variations of SUVmax by response : 8 partial response and 2 stable disease
Measure: Median (Standard Deviation); unit: change in relative variance
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
change in relative variance
  Partial response: number analyzed (Participants) | 8
  Partial response | 38.6 (274.5)
  Stable disease: number analyzed (Participants) | 2
  Stable disease | -18.0 (40.1)
Statistical Analysis 1: Comparison: Functional Imaging; Test type: Superiority — alpha=5%; p = 0.192, Kruskal-Wallis; Mean Difference (Net) = 1.705

53. Secondary Outcome: Peritoneal Extent Assessed by Fagotti Score Using MRI Data
Description: The Fagotti score ranges from 0 to 14 and is used to evaluate the peritoneal damage of patients. This score was collected during pretherapy and after 4 cycles of chemotherapy. The higher the stage number is, the further the cancer has spread.
  The Fagotti questionnaire has 7 items. A subscale value of 0 or 2 is assigned depending on whether the disease is present in those specific sites : large omentum, peritoneal carcinosis , diaphragmatic carcinosis, mesenteric retraction, intestinal infiltration, stomach infiltration,liver metastases.
  The sum of subscale values corresponds to Fagotti score.
Time Frame: Pre-therapeutic
Measure: Count of Participants; unit: Participants
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
Participants
  4 | 2
  8 | 4
  10 | 2
  12 | 1
  Missing | 1

54. Secondary Outcome: Peritoneal Extent Assessed by Fagotti Score Using MRI Data
Description: TThe Fagotti score ranges from 0 to 14 and is used to evaluate the peritoneal damage of patients. This score was collected during pretherapy and after 4 cycles of chemotherapy. The higher the stage number is, the further the cancer has spread.
  The Fagotti questionnaire has 7 items. A subscale value of 0 or 2 is assigned depending on whether the disease is present in those specific sites : large omentum, peritoneal carcinosis , diaphragmatic carcinosis, mesenteric retraction, intestinal infiltration, stomach infiltration,liver metastases.
  The sum of subscales corresponds to Fagotti score.
Time Frame: Interval surgery visit: up to 3 weeks after cycle 4 of chemotherapy and until the day before the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
Participants
  0 | 1
  2 | 1
  4 | 2
  6 | 2
  8 | 3
  10 | 1

55. Secondary Outcome: Overall Survival
Time Frame: 10 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
percentage of patients | 90 [47.3 to 98.5]

56. Secondary Outcome: Progression-free Survival as Per RECIST v1.1
Time Frame: 9, 13, 14 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Functional Imaging
Number analyzed (Participants) | 10
percentage of patients
  9 months | 90.0 [47.3 to 98.5]
  13 months | 78.8 [38.1 to 94.3]
  14 months | 67.5 [29.1 to 88.2]

ADVERSE EVENTS:
Time Frame: All adverse events are recorded from the first visit (J0 inclusion) until 4 weeks after the third PET/MRI examination. Beyond this period, only SAE likely to be related to the research or the medical device or to the procedure of implementation of the medical device are reported.
Arm/Group | Functional Imaging
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Imaging (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1) — Blood and lymphatic system disorders
Colonic obstruction (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders
Vomiting (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders
Sepsis (Infections and infestations) | 1 (1) — Infections and infestations
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Imaging (N=11)
Anemia (Blood and lymphatic system disorders) | 3 (3) — Blood and lymphatic system disorders
Sinus tachycardia (Cardiac disorders) | 1 (1) — Cardiac disorders
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders
Ascites (Gastrointestinal disorders) | 2 (2) — Gastrointestinal disorders
Bloating (Gastrointestinal disorders) | 1 (1) — Gastrointestinal disorders
Constipation (Gastrointestinal disorders) | 2 (2) — Gastrointestinal disorders
Diarrhea (Gastrointestinal disorders) | 2 (2) — Gastrointestinal disorders
Nausea (Gastrointestinal disorders) | 2 (2) — Gastrointestinal disorders
Fatigue (General disorders) | 2 (2) — General disorders and administration site conditions
Fever (General disorders) | 2 (2) — General disorders and administration site conditions
Allergic reaction (Immune system disorders) | 2 (4) — Immune system disorders
Bronchial infection (Infections and infestations) | 2 (2) — Infections and infestations
Enterocolitis infectious (Infections and infestations) | 1 (1) — Infections and infestations
Peritoneal infection (Infections and infestations) | 1 (1) — Infections and infestations
Urinary tract infection (Infections and infestations) | 2 (2) — Infections and infestations
Creatinine increased (Investigations) | 1 (1) — Investigations
Neutrophil count decreased (Investigations) | 1 (1) — Investigations
Platelet count decreased (Investigations) | 1 (1) — Investigations
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Musculoskeletal and connective tissue disorders
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Musculoskeletal and connective tissue disorders
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) — Nervous system disorders
Cystitis noninfective (Renal and urinary disorders) | 1 (1) — Renal and urinary disorders
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2) — Renal and urinary disorders
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) — Reproductive system and breast disorders
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) — Reproductive system and breast disorders
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory, thoracic and mediastinal disorders
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) — Skin and subcutaneous tissue disorders
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) — Skin and subcutaneous tissue disorders
Hypertension (Vascular disorders) | 2 (2) — Vascular disorders
Thromboembolic event (Vascular disorders) | 1 (1) — Vascular disorders

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes